CLINICAL TRIAL: NCT04313205
Title: A Randomized, Open-label, Multiple-dose, Two-period, Crossover, Study to Investigate the Pharmacokinetic Profile of 2 Formulations of JKB-122 in Healthy Male Subjects
Brief Title: A Pharmacokinetic Study of JKB-122 Tablets Compared to Capsule
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: TaiwanJ Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TWJ-SR122
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Autoimmune Hepatitis
MeSH Terms: conditions — Hepatitis, Autoimmune | interventions — JKB-122; Capsules

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Capsule (Active Comparator): JKB-122 capsule on period 1 followed by JKB-122 Tablet on period 2
  Interventions: Drug: JKB-122 in capsule or tablet form
- Tablet (Active Comparator): JKB-122 tablet on period 1 followed by JKB-122 capsule on period 2
  Interventions: Drug: JKB-122 in capsule or tablet form

INTERVENTIONS:
Drug: JKB-122 in capsule or tablet form — JKB-122 is a TLR4 antagonist and will be administrated in capsule or tablet form

SUMMARY:
The purpose of this study is to compare the pharmacokinetics of JKB-122 tablets with JKB-122 capsules in healthy male subjects subjects.

DETAILED DESCRIPTION:
This clinical study will be a randomized, open-label, multiple-dose, two-period, crossover study in healthy male subjects. After screening, subjects will be randomized to receive either JKB-122 tablet or JKB-122 capsule in a 1:1 ratio. There will be two dosing periods (Period 1 and Period 2). Subjects who receive JKB-122 capsule during Period 1 will receive JKB-122 tablet during Period 2 and vice versa. The 2 dosing periods will be separated by a washout period.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has a body mass index (BMI) range of 18.5 and < 25.0 kg/m2 and weighs at least 50 kg.
2. Agreement for subject and female partner of childbearing potential to use acceptable method of contraception
3. The subject provided written informed consent.

Exclusion Criteria:

1. Any history or evidence of any clinically significant major disease or malignancy, as judged by the Investigator.
2. Any clinically significant abnormality following the Investigator's review of the physical examination, ECG and clinical study protocol-defined clinical laboratory tests.
3. Use of prescribed or non-prescribed drugs (including vitamins, natural and herbal remedies, e.g. St. John's Wort) in the 2 weeks prior to study drug administration.
4. Consumption of grapefruit, pomelo, citrus fruits, starfruit, pomegranate, papaya, mango, rambutan, kiwi fruit, dragon fruit or passion fruit and products containing these fruits in the 2 weeks prior to study drug administration.
5. Current smoker or history of smoking within 3 months before the Screening Visit.
6. History of drinking more than 21 units of alcohol per week within 3 months prior to the Screening Visit.
7. Any use of drugs-of-abuse within 3 months before the Screening Visit.
8. Any significant blood loss or donation of blood (250 ml within 2 months or 500 ml within 3 months) prior to study drug administration.
9. Positive serology test for hepatitis B surface antigen (HBsAg), hepatitis C virus antibodies (HCVAb) or human immunodeficiency virus.
10. Participation in any clinical study or administration of any investigational product within 1 month of study drug administration.
11. The subject has any other condition, which in the opinion of the Investigator precludes the subject's participation in the clinical study.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Area under the curve from the time of dosing to steady state (AUC¬(0-τ)ss¬¬) | 2 WEEKS
  Plasma PK parameters will be measured comparison between JKB-122 capsule and JKB-122 tablet

SECONDARY OUTCOMES:
Number of Adverse events (AEs) observed | 2 WEEKS
  Safety observation of the drug treatment.

IPD SHARING:
Plan to Share IPD: No